CLINICAL TRIAL: NCT06029959
Title: Optimizing Adherence to the Treatment of Sleep Apnea Among Patients With Stroke Undergoing Inpatient Rehabilitation
Brief Title: Stroke and CPAP Outcome Study 3
Acronym: SCOUTS3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sandeep Khot, Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016907; 1R01HL164394-01A1 (NIH)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke; Intra Cerebral Hemorrhage; Obstructive Sleep Apnea; Adherence, Treatment; Motivation
Keywords: behavioral therapy; continuous positive airway pressure; rehabilitation therapy; stroke recovery; self determination
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Sleep Apnea, Obstructive; Treatment Adherence and Compliance | interventions — Continuous Positive Airway Pressure; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SCOUTS3 Optimization Arm (Experimental): In a single-arm study, participants from acute ischemic stroke or intraparenchymal hemorrhage within the past 30 days will be tested for OSA with a single-night portable OSA test during inpatient rehabilitation (IPR). Eligible participants will then be started on continuous positive airway pressure (CPAP) therapy and exposed to a multicomponent CPAP adherence intervention, beginning during IPR and extending for 3 months. Participants' CPAP use will be monitored, and input regarding the intervention will be sought from the participants, CPAP partners, and the research team implementing the intervention. Data from an initial group of study participants will be reviewed in meetings with the study team and a patient advisory board, and adaptations will be devised and then implemented within the next batch of study participants. Through this iterative process that includes input from important stakeholders, the behavioral intervention will be adapted for use among stroke patients.
  Interventions: Device: Continuous positive airway pressure (CPAP); Behavioral: CPAP technical support intervention; Behavioral: Motivational Enhancement Therapy (MET); Behavioral: Mobile Health intervention

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Eligible participants with a diagnosis of OSA will be set up with autotitrating CPAP by the study's sleep technologist. The CPAP device includes an auto-titrator that adjusts the delivered pressure between 5 to 15 cm of water to eliminate obstructive events.
Behavioral: CPAP technical support intervention — SCOUTS 3 sleep technologists (ST) will make mask type/size or device adjustments, as needed, and provide training to participants and CPAP partners to improve skills involved with mask placement and device maintenance. For participants with non-acceptance of CPAP over the first night, a standardized desensitization program will be implemented. Persistent problems with CPAP use or mask fit, or any high residual respiratory events will be discussed between the sleep technologist and the study's board-certified sleep medicine physician.
Behavioral: Motivational Enhancement Therapy (MET) — In-person Motivational Enhancement Therapy (MET) sessions by a trained sleep coach will occur within a week of starting CPAP and, with permission, conducted with a CPAP partner, when available. The MET session recordings will be uploaded into the HIPAA compliant Lyssn platform for evaluation, including feedback to the sleep coach. The goal will be 5 total MET sessions, either in-person or by phone, spanning the inpatient and then outpatient settings.
Behavioral: Mobile Health intervention — Study participants will be assisted in registering for and trained on the ResMed myAir app. Participants will also receive mobile health messages based on Self-Determination Theory.

SUMMARY:
A problem with breathing during sleep, called obstructive sleep apnea (OSA), likely increases the risk of stroke and is common in people who have had a stroke, present in about 2/3 of stroke survivors. There is also evidence that OSA predicts worse outcome after stroke. The question being addressed in the Stroke and CPAP Outcome Study 3 (SCOUTS3) is how to improve use of continuous positive airway pressure (CPAP) therapy to treat OSA when started during intensive stroke rehabilitation.

DETAILED DESCRIPTION:
In an initial single-arm study, participants with stroke will be tested for OSA and treated with auto-titrating CPAP during inpatient stroke rehabilitation and continued for a 3-month treatment period. Multiple behavioral interventions will be used to improve CPAP use, including intensive CPAP technical support, motivational enhancement therapy, and phone and mobile health automated support. The multicomponent behavioral intervention will be optimized to improve CPAP adherence with the engagement and input of stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Head CT or brain MRI demonstrating an acute ischemic infarction or intraparenchymal hemorrhage within past 30 days
* Person providing consent (patient or legally authorized representative) able to be consented in English or Spanish

Exclusion Criteria:

* Unable to obtain informed consent from participant or surrogate
* Incarcerated
* Known pregnancy
* Current mechanical ventilation, tracheostomy or supplemental oxygen use > 4L/min
* Current use of positive airway pressure or use within 14 days prior to stroke
* History of pneumothorax, bullous emphysema or other serious co-morbid conditions which limit CPAP use
* Stroke related to tumors, vascular malformations or subarachnoid hemorrhage
* Active use of sedative drugs that can interfere with testing for obstructive sleep apnea (OSA)
* Anticipated inpatient rehabilitation length of stay < 3 nights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Khot, MD, MPH, Principal Investigator — University of Washington; Devin Brown, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: NIH Reporter — http://reporter.nih.gov/search/b05ZXayvqUCz6wIm20U-rw/project-details/10658404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2023 and September 2024, 36 IPR patients with ischemic stroke or intracerebral hemorrhage were enrolled.
Pre-assignment Details: A single-night portable sleep apnea test was performed at a mean of 16.0 days from stroke onset and 4.0 days from IPR admission.
Period: Overall Study
Arm/Group | SCOUTS3 Optimization Arm
Started | 36
Completed | 30
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | SCOUTS3 Optimization Arm
Number analyzed (Participants) | 36
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 56.7 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 7
  Unknown or Not Reported | 0
Respiratory event index (REI) [Mean (Standard Deviation); unit: events per hour] — Number of respiratory events (apneas and hypopneas) per hour
  events per hour | 21.3 (14.7)
Oxygen desaturation index (ODI) [Mean (Standard Deviation); unit: events per hour] | 18.1 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: CPAP Adherence
Description: Mean hours of nightly CPAP use during and after inpatient rehabilitation over 3 months
Time Frame: From CPAP initiation after study enrollment and sleep apnea testing to 90 days from CPAP initiation
Measure: Mean (Standard Deviation); unit: nightly hours of CPAP use
Arm/Group | SCOUTS3 Optimization Arm
Number analyzed (Participants) | 30
nightly hours of CPAP use | 3.1 (2.6)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- SCOUTS3 Optimization Arm: In a single-arm study, participants with ischemic stroke or intraparenchymal hemorrhage within 30 days will be tested for obstructive sleep apnea with a portable test during inpatient rehabilitation (IPR). Eligible participants will be started on autotitrating continuous positive airway pressure (CPAP) therapy and exposed to a multicomponent adherence intervention, beginning during IPR and extending for 3 months. Input regarding the intervention will be sought from the participants, CPAP partners, and the research team implementing the intervention. Data from an initial group of participants will be reviewed, and adaptations will be implemented within the next batch of participants. Through this iterative process, the behavioral intervention will be adapted for use among stroke patients.
  CPAP technical support intervention: SCOUTS 3 sleep technologists will make mask type/size or device adjustments, as needed, and provide training to participants and CPAP partners to improve skills involved with mask placement and device maintenance.
  Motivational Enhancement Therapy (MET): In-person Motivational Enhancement Therapy sessions by a trained sleep coach will occur within a week of starting CPAP and, with permission, conducted with a CPAP partner.
  Mobile Health intervention: Study participants will be assisted in registering for and trained on the ResMed myAir app. Participants will also receive mobile health messages based on Self-Determination Theory.
Arm/Group | SCOUTS3 Optimization Arm
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT06029959/Prot_SAP_001.pdf